CLINICAL TRIAL: NCT06777797
Title: Prospective, Verification Study to Assess Condom Fit Across Polyurethane (PU) and Natural Rubber Latex (NRL) Condoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5068701
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Condom Use

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, intra-individual, exploratory, single-centre clinical investigation. Each participant will test 4 PU condoms and 4 NRL condoms in a defined order, according to the randomization schedule.
Masking Description: Although it is an open label investigation, some information such as condom size will be removed from all packages so participants will not know which condom variant they are testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PU condom (Experimental): Following randomization, participants will test PU condoms first followed by NRL condoms.
  Interventions: Device: PU condoms (Test PU Condom A, Test PU Condom B, Test PU Condom C, Test PU Condom D)
- NRL condom (Experimental): Following randomization, participants will test NRL condoms first followed by PU condoms.
  Interventions: Device: NRL condoms (Test NRL Condom A, Test NRL Condom B, Test NRL Condom C, Test NRL Condom D)

INTERVENTIONS:
Device: PU condoms (Test PU Condom A, Test PU Condom B, Test PU Condom C, Test PU Condom D) — Participants will be provided with PU condoms (2 condoms per variant) to use during masturbation.
  Arms: PU condom
Device: NRL condoms (Test NRL Condom A, Test NRL Condom B, Test NRL Condom C, Test NRL Condom D) — Participants will be provided with NRL condoms (2 condoms per variant) to use during masturbation.
  Arms: NRL condom

SUMMARY:
The investigation is to explore condom experience in terms of comfort and fit across a range of condom sizes and materials.

DETAILED DESCRIPTION:
In this investigation, 4 Polyurethane (PU) condom variants and 4 Natural Rubber Latex (NRL) condom variants will be tested by participants to explore condom experience.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before participation in the clinical investigation.
2. Cisgender male, aged 18 - 55 years.
3. In the opinion of Investigator, experienced user of condoms who use condoms to prevent pregnancies and / or contracting STIs.
4. Able and willing to achieve a penile erection following self-stimulation.
5. Able and willing to masturbate with a PU or NRL condom on.
6. Agree to use only lubricant provided by the study for use with IMDs, if required.
7. Agree not to wear any genital piercing jewelry while using the study condoms.
8. Agree not to use sex toys, consume alcohol or use drugs intended to enhance or diminish sexual response when using study condoms.
9. Agree to perform erected penis size measurement at site and at home.

Key Exclusion Criteria:

1. Participants with known trouble attaining or maintaining an erection.
2. Participants presenting clinically abnormal findings on the penis that in the opinion of the investigator can affect the study outcome.
3. Participants with an allergy or sensitivity to the ingredients of the test products, including the test condoms or any lubrication products provided.
4. Use of any topical medications applied to the penis between screening and visit 3.
5. Participants with diagnosed or suspected erectile dysfunction.
6. Participants with a history of prostatectomy.
7. Participants with a history of urethral surgery.
8. Participants with any other congenital or acquired genital abnormalities (e.g. peyronies disease, hypospadias, intersex, phimosis, penile cancer).
9. Psychiatric conditions that might limit the participation in the clinical investigation and/or that lead to the assumption that the ability to completely understand the consequences of consent is missing.
10. Participants with any medical condition in the opinion of the investigator which poses a risk to the participant or is detrimental to the objectives of the clinical investigation.
11. Participants who should not participate in the clinical investigation for any other reason as judged by the investigator.
12. Participation in a pharmaceutical trial with investigational products or in a clinical investigation with another medical device within the last 30 days prior to the visit 2 (day 1) and / or during this clinical investigation.
13. Employees of the investigation sites who are directly involved in this clinical investigation or employees of the sponsor's company.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender male
Enrollment: 224 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
The exploration of condom experience across a range of sizes and materials | 6 weeks condom use period (intervention duration)
  Participants will measure their penis size at screening and will be assigned to pre-defined groups. The endpoint is the exploration of condom experience across a range of materials and sizes within each group. Participants will evaluate the condoms over a period of 6 weeks and rate their condom experience through subject perceived questionnaires using the following scales:
  1. Disagree, somewhat disagree, neither agree nor disagree, agree, strongly agree;
  2. 1-10 with 1 being extremely dissatisfied and 10 being extremely satisfied.

SECONDARY OUTCOMES:
Examine whether the preferred condom variant is the same for both PU and NRL condoms. | 6 weeks condom use period (intervention duration)
  The endpoint is the evaluation of the correspondence of preferred condom variant for PU and NRL condoms. The endpoint is collected over a period of 6 weeks on different condom types and variants by means of subject perceived questionnaires which participants will rate their condom preference using the following scales:
  1. Disagree, somewhat disagree, neither agree nor disagree, agree, strongly agree;
  2. 1-10 with 1 being extremely dissatisfied and 10 being extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as per local regulations.